CLINICAL TRIAL: NCT06352034
Title: Effectiveness of Empathy Training Among Psychology Students Trainees: A Randomized Controlled Trial
Brief Title: Empathy Training for Psychology Students Trainees
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Empathy Training for Students
Record Dates: First submitted 2024-03-21; First posted 2024-04-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Empathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empathy Training (Experimental): The Empathy training consists of five sessions. Each session contains psychoeducation, three-role group exercises, and Q&A. The interval between every session is 5-14 days. Sessions are scheduled for 1.5 hours, including 30 minutes of psychoeducation, 45 minutes of three-role group exercises, and 15 minutes of Q&A.
  Interventions: Behavioral: Empathy Training
- Wait-List (No Intervention): The participants in the wait-list group will not receive the empathy training or other similar training until all the groups finish their one-month follow-up measurements.

INTERVENTIONS:
Behavioral: Empathy Training — The intervention contains five themes: 1) An overview of empathy and emotions. 2) Cognitive empathy and clarification technique. 3) Emotional empathy and reflection of feelings technique. 4) Awaring and dealing with the inner feelings while empathizing. 5) Empathy timing and "emotional pendulum" technique.
  Arms: Empathy Training

SUMMARY:
This study aims to examine the effectiveness of empathy training for psychology student trainees who plan to become mental health practitioners. The training consists of five sessions of psychoeducation, three-role group exercises, and Q&A. Empathy assessment will be based on self-reported, listener-reported, and observer-reported measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female (aged between 18 and 65 years old)
* Major or double major in psychology
* Currently enrolled undergraduate or graduate students
* Taking psychological counselor as one of the major occupational chooses

Exclusion Criteria:

* Hearing, speech, reading, or writing impairments
* A diagnosis of mental disorders
* Simultaneously participating in other emotional skills training
* Suicidal ideation or self-injurious behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from counseling duration | Through study completion, an average of 3 month
  A 10-minute counseling simulation will be conducted for each participant. The simulation will last 10 minutes or before 10 minutes if the participant gives up midway. The duration time will be recorded to measure the counseling tolerance of the participants. Longer duration indicates better counseling tolerance.
Change from Baseline of 12-Item Version of the Barrett-Lennard Relationship Inventory | Through study completion, an average of 3 month
  A 12-item empathy self-report, senior-psychological-counselor-report, and simulate-client-report scale measures regard (R), empathic understanding (E), congruence (C), and unconditionality of regard (U) of the therapist. The scoring of each item is from -3 to +3 (12 items, total score varies from -36 to 36). A higher score represents better facilitative conditions the therapist can shape.
Change from consultation willingness question inquiry | Through study completion, an average of 3 month
  A single item inquiry "How willing are you to come back for consultation next time?" will be asked to the simulation "client" to measure the ability to build the counselor-client relationship. The item scores from 0 to 4. A higher score represents a higher ability to build the counselor-client relationship.
Change from morphed emotion perception task | Through study completion, an average of 3 month
  An experimental task measures the ability of emotion perception. Participants need to identify the emotion of facial pictures out of six basic emotions (i.e., anger, sadness, fear, disgust, surprise, and happiness). The higher accuracy indicates better emotion perception ability.
Change from Baseline of the Measure of Empathy Scale | Through study completion, an average of 3 month
  An 8-item empathy self-report scale measures cognitive empathy and emotional empathy on a 5-point Likert scale (score from 1 to 5, and total score vary from 8 to 40). A higher score represents higher empathy ability.
Change from Baseline of the Emotion Perception Scale | 1 month
  A 13-item emotion perception scale measures the extent of emotions within a month, including anger, happiness, sadness, fear, surprise, disgust, guilt, shame, pressure, depression, inner anger, numbness, and aggrievedness. Each item scores from 0 to 5, with total score varying from 0 to 65. A higher score represents a higher extent of feeling the emotions.
Change from Baseline of the Peking Alexithymia Scale | 1 month
  A 23-item Peking alexithymia scale measures the ability and willingness to feel, recognize, and share emotions on a 5-point Likert scale (scores from 1 to 5, and total scores vary from 23 to 115). A higher score represents more severe alexithymia.

SECONDARY OUTCOMES:
Change from Baseline of the Patient Health Questionnaire | 2 weeks
  The 9-item patient health questionnaire (PHQ-9) measures the depression symptoms (scores from 0 to 3, and total score vary from 0 to 27). A higher score represents worse depression symptoms.
Change from Baseline of the Generalized Anxiety Disorder Scale | 2 weeks
  The generalized anxiety disorder-7 scale (GAD-7) measures the generalized anxiety disorder symptoms (scored from 0 to 3, and total score from 0 to 21). A higher score represents worse anxiety symptoms.
Change from Baseline of the Peking Irritability Scale | 1 month
  A 17-item irritability measurement scale, Peking irritability scale, measures impulsive emotions, thoughts, and behaviors on a 5-point Likert scale (score from 1 to 5, and total score vary from 17 to 85). A higher score represents higher irritability.
Change from Baseline of the the Fatigue Assessment Scale | Through study completion, an average of 3 month
  A 10-item fatigue assessment scale measures the degree of fatigue (score from 1 to 5, and total score vary from 10 to 50). A higher score represents a higher degree of fatigue.
Change from Baseline of the the Patient Health Questionnaire | 4 weeks
  A 21-item patient health questionnaire measures the extent of semantic symptoms (score from 0 to 2, and total score vary from 0 to 42). A higher score represents a higher degree of semantic problems.
Change from Baseline of the Cognitive-Emotion Regulation Questionnaire | Through study completion, an average of 3 month
  An 18-item cognitive-emotion regulation questionnaire measures regulation strategy (score from 1 to 5, and total score vary from 18 to 90). A higher score represents higher cognitive-emotion regulation ability.
Change from Baseline of the Difficulties in Emotion Regulation Scale | Through study completion, an average of 3 month
  A 36-item difficulties in emotion regulation scale measures emotion regulation difficulties (score from 1 to 5, and total score vary from 36 to 180). A higher score represents higher difficulties in emotion regulation.
Change from Baseline of the the Satisfaction with Life Scale | Through study completion, an average of 3 month
  A 5-item satisfaction with life scale measures life satisfaction (score from 1 to 7, and total score vary from 5 to 35). A higher score represents more satisfaction with life.
Change from Baseline of the the Subjective Happiness Scale | Through study completion, an average of 3 month
  A 4-item subjective happiness scale measures happiness (score from 1 to 7, and total score vary from 4 to 28). A higher score represents a happier state.
Change from Baseline of the Connor-Davidson Resilience Scale | 1 month
  A 10-item Connor-Davidson resilience scale measures resilience (score from 0 to 4, and total score vary from 0 to 40). A higher score represents a higher degree of resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Yinyin Zang, PhD, Principal Investigator — Study Principal Investigator Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China